CLINICAL TRIAL: NCT07245615
Title: The Effects of Different Vibro-tactile Stimulation Intensities on Head Posture in Cervical Dystonia
Brief Title: Effect of Vibro-tactile Stimulation Intensity on Head Posture in Cervical Dystonia
Acronym: (CD-VTS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00024537
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Cervical Dystonia
Keywords: vibrotactile stimulation; non-invasive; symptom control; proprioception
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Dystonia Group (Experimental): All participants with cervical dystonia will be in this group to receive the intervention. After answer three questionnaires (The Mini Mental State Examination, the Revised Toronto Western Spasmodic Torticollis Rating Scale and Psychiatric Screening Tool, Fahn, Tolosa, Marin Tremor Rating Scale), their neck, wrist, and ankle proprioception will be tested respectively. They they will go through the intervention of cervical vibrotactile stimulation. Lastly, their neck proprioception will be tested again.
  Interventions: Device: cervical vibrotactile stimulation
- Healthy Controls (No Intervention): Healthy people age- and sex- matched with participants with cervical dystonia will be in this group. This group will only be tested on their neck, wrist, and ankle proprioception, to compare with the cervical dystonia group.

INTERVENTIONS:
Device: cervical vibrotactile stimulation — The intervention in this study is vibrotactile stimulation with 3 different intensities on 4 combinations of cervical muscles. The three intensity levels are 0.25mm, 0.64mm, and 1.48mm of movement range of the vibrator, when attached to the cervical area. The four muscle combinations (left and right SCM, left and right TRP, left SCM and TRP, right SCM and TRP) are selected as they were shown to be more effective than other combinations in a previous studies. The total number of bouts of stimulation is 12 (3 intensities * 4 muscle combinations). Each VTS application is 2 minutes long, resulting in total stimulation time of 24 minutes. There will be a 5-minute break of no-vibration between each application of vibration.
  During the intervention, the participant will remain seated and asked to not interfere voluntarily with dystonic muscle spasms. During breaks, they can adjust their head posture for their comfort. Extra breaks will be given if needed.
  Arms: Cervical Dystonia Group

SUMMARY:
The primary goal of this clinical trial is to examine the effects of cervical vibrotactile stimulation intensity on abnormal head posture in people with cervical dystonia. The main question is: Does higher vibration intensity correct head posture to a greater extent than lower vibration intensity? Researchers will compare the head posture of participants with cervical dystonia who receive different intensities of vibration to cervical muscles.

The secondary goal of this clinical trial is to examine the degree of proprioceptive impairment in cervical dystonia. Specifically, the study will assess proprioceptive impairment at the neck, wrist, and ankle joints, and seeks to determine whether the impairment improves with cervical vibrotactile stimulation.

Researchers will compare the proprioception testing results of these joints between cervical dystonia patients and age- and sex- matched healthy controls. Researchers will also compare the neck proprioception testing results of cervical dystonia patients before and after stimulation.

Participants will visit the lab once for three hours, where they will go through:

1. clinical questionnaires;
2. neck, wrist, and ankle proprioception testing,
3. vibrotactile stimulation where they sit and relax
4. neck proprioception testing

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of adult-onset, isolated idiopathic cervical dystonia.

Exclusion Criteria:

History of other neurological diseases, including Parkinson's disease, essential tremor, dementia, etc.

History of peripheral nervous system disease that can impair proprioception. Deep brain stimulation implanted or denervation surgery. UBACC score lower than 15. Severe head tremors or facial muscle contractions. Regular intake of benzodiazepines or antidepressant medication.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Head Angle Index | As part of the one-time visit, this part will take 90 minutes.
  The primary outcome measure is the head angle index, which quantifies how much a participant's head posture deviates from a neutral upright position. There are three degrees of freedom for the neck joint (axial rotation, lateral bending, and flexion/extension). For each participant, the degree(s) of freedom with abnormality will be identified at baseline. For any time period during the experiment, the mean absolute neck angle in each abnormal degree of freedom will be calculated and normalized by the typical maximal range of motion in healthy individuals. These normalized values will be averaged to yield the Head Angle Index.

SECONDARY OUTCOMES:
Position Matching Error | As part of the one-time visit, this part will take 60 minutes.
  The secondary outcome measure is absolute position matching error, which quantifies the position sense acuity of the participants in each joint. For each tested joint, they will be given a set of target position. The joint will be passively rotated to the target position, and back to the starting position. The participant will then try to reproduce the target position, based on their memory of the position. After repeating for 9 times, the absolute value of the differences between the matched position and the target position will be averaged to get the absolute position matching error.
the Toronto Western Spasmodic Torticollis Rating Scale Score | As part of this one-time visit, 10 minutes.
  This three-part rating scale will evaluate the severity, disability and pain level of each CD participant. Each part results in a numerical score.
Fahn-Tolosa-Marin Clinical Rating Scale Score | As part of a one-time visit, 10 minutes.
  Tremor severity level will be evaluated with this numerical score.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Sensorimotor Control Laboratory, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No